CLINICAL TRIAL: NCT02923804
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of MF4637 for Correcting the Omega-3 Nutritional Deficiency in NAFLD Patients When Added to Standard of Care
Brief Title: Evaluation of MF4637 for Correcting the Omega-3 Nutritional Deficiency in NAFLD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1051-001-PRO-19012015
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2016-09

CONDITIONS: Non Alcoholic Fatty Liver
Keywords: steatosis; NAFL; NAFLD; Polyunsaturated fatty acids; omega-3; EPA; DHA; fish oil
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Experimental): 3 capsules of 1g concentrated omega-3 taken daily for 6 months
  Interventions: Dietary Supplement: Omega-3
- Olive oil (Placebo Comparator): 3 capsules of 1g olive oil taken daily for 6 months
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Omega-3 — 3x 1g capsules taken daily for 6 months
  Arms: Omega-3
Dietary Supplement: Olive oil — 3x 1g capsules taken daily for 6 months
  Arms: Olive oil

SUMMARY:
This study is a prospective, randomized, placebo-controlled, double-blind trial to determine the effect of high concentrate omega-3 capsules on the omega-3 status of patients with non-alcoholic fatty liver.

DETAILED DESCRIPTION:
Subjects with non-alcoholic fatty liver (simple steatosis) confirmed within the last year by ultrasound or other imaging modality will be recruited to the study. Subjects will be randomized to a treatment arm of high concentrate capsules or placebo for a 6 month treatment period.Omega-3 content of red blood cells (omega-3 index) will be measured for primary endpoint assessment. Quantitative MRI will be performed to determine the effect on liver fat content.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history of clinical diagnosis of NAFLD by ultrasound, MRI or biopsy within one (1) year prior to screening (V1). If the diagnostic test date is greater than one (1) year, abdominal ultrasound will be repeated at (V1) and must confirm a diagnosis of NAFLD.
2. Men or women, ≥18 years of age.
3. BMI between 18.0 and 39.9 kg/m2.
4. Non-smokers (>3 months of non-smoking).
5. If on a statin regimen, history (> 1 month stable dose) of taking a statin medication (HMG-CoA reductase inhibitor example: Lipitor, Zocor, Crestor, Pravachol, Lescol, Livalo, etc).
6. Able to understand and cooperate with study procedures, and have signed a written informed consent prior to any study procedures.

Exclusion Criteria:

1. Diagnosis of NASH.
2. Bilirubin >2x ULN.
3. Other causes of liver inflammation including Hepatitis A, B or C, HIV, confirmed or suspected cirrhosis, Wilson's disease, autoimmune hepatitis, hemochromatosis, alcoholic steatohepatitis, pancreatitis, or prescription medications known to cause liver damage, or known to be hepatotoxic.
4. Subjects with a history of bariatric surgery.
5. Significant weight loss (> 5% body weight) or rapid weight loss (>1.6 kg/week), within six months of screening.
6. Current or recent (within six months of screening) history of significant gastrointestinal, renal, pulmonary, hepatic or biliary disease, endocrine diseases or other invasive weight loss treatments (Type II Diabetes permitted, and stable (> 3 months) thyroid disorders).
7. Individual taking prescription or over-the-counter medications (including dietary supplements, see Appendix 1) known to alter lipid metabolism, within four (4) weeks of randomization. These medications include (but are not limited to) the following: bile acid sequestrants, cholesterol absorption inhibitors, niacin or fibrates,
8. Individuals taking prescription omega-3 fatty acids.
9. Use of supplements including Omega-3s and Omega-6s, other oil-based supplements, phytosterols, Vitamin E, prebiotics and probiotics, or any weight loss supplements within four (4) weeks of randomization (multivitamins and minerals containing Vitamin E are permitted).
10. Use of systemic corticosteroids, androgens (except androgens for hypogonadism to restore normal levels), phenytoin, erythromycin and other macrolides, thiazolidinediones (e.g. pioglitazone), and thyroid hormones (except stable-dose thyroid replacement therapy for four (4) weeks prior to enrollment).
11. Use of the anticoagulants warfarin (Coumadin), dabigatran (Pradaxa), apixaban (Eliquis) or rivaroxaban (Xarelto). NOTE: Anti-platelet agents such as Plavix are allowed.
12. Pregnant or lactating women or women of childbearing potential, who are not using an approved method of contraception. A woman is considered to be of childbearing potential unless she is post-hysterectomy, one or more years postmenopausal, or one or more years post-tubal ligation.
13. History of significant cardiovascular or coronary heart disease (CVD or CHD) as defined by having had a coronary artery bypass procedure, coronary stent or angioplasty, or myocardial infarction in the previous six (6) months.
14. History of cancer, other than non-melanoma skin cancer and basal cell carcinoma, within the previous five years.
15. Poorly controlled or uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥95 mmHg).
16. Recent history of prolonged alcohol (>3 months) use (within past 6 months) or excessive alcohol use, defined as >14 drinks per week (one drink = 12 oz. beer, 4 oz. wine, 1.5 oz. hard liquor).
17. Exposure to any investigational agent within four (4) weeks prior to Visit 1.
18. Subjects planning to undergo surgery during the study period or up to 1 month after the study
19. Any serious psychiatric disease or disorder, which, in the opinion of the investigator, would preclude the subject from participating in the study.
20. Any known intolerance to the investigational ingredients of this medical food.
21. Has a condition the Investigator believes would interfere with the evaluation of the subject, or may put the subject at undue risk during the course of the study, including potentially abnormal lab results, due to a traumatic event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
• The primary endpoint is the difference in mean percent changes from baseline (Week 24 each with baseline subtracted) between placebo and omega-3 groups | 6 months

SECONDARY OUTCOMES:
• Difference in mean percent change from baseline to end-of-treatment in RBC EPA and RBC DHA (percentage of lipids and quantitative measurements) | 6 months
• Difference in mean percent change from baseline to end of treatment in omega-6: omega-3 ratios. | 6 months
To assess the impact of omega-3 on changes in liver fat as determined by MRI-PDFF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Derek Tobin, PhD, Study Director — BASF
Locations (6):
- United States (6):
  - Hialeah, Hialeah, Florida
  - Lake Worth, Lake Worth, Florida
  - Lauderdale Lakes, Lauderdale Lakes, Florida
  - Miami, Miami, Florida
  - Greenville, Greenville, South Carolina
  - Arlington, Arlington, Texas

IPD SHARING:
Plan to Share IPD: No